CLINICAL TRIAL: NCT05508451
Title: Comparison of the Efficacy of Tenoxicam, Paracetamol (Acetaminophen), and Tenoxicam-Paracetamol Combination on Postoperative Pain in Double-Jaw Surgery Patients
Brief Title: Comparison of the Effects of Tenoxicam and Paracetamol on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, seher orbay yasli, Medical Doctor, Anesthesiologist, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/303
Record Dates: First submitted 2022-08-13; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Pain, Acute
Keywords: Maxillofacial Orthognathic Surgery; Pain management; Postoperative pain; Tenoxicam
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- paracetamol (Active Comparator)
  Interventions: Procedure: Double jaw surgery
- tenoxicam (Active Comparator)
  Interventions: Procedure: Double jaw surgery
- tenoxicam+paracetamol (Active Comparator)
  Interventions: Procedure: Double jaw surgery
- placebo (Placebo Comparator)
  Interventions: Procedure: Double jaw surgery

INTERVENTIONS:
Procedure: Double jaw surgery — A type of orthognathic surgery

SUMMARY:
Postoperative pain is generally caused by inflammation and oedema related to tissue trauma. Surgical tissue trauma is caused by many factors such as cotery-related burns, surgical incisions, dissections, and instrumental procedures like cutting, stretching, or compression.

The pain stimulus is triggered by mediators released by the traumatic tissue and transmitted to the spinal cord and then to the upper centres of the brain. Tenoxicam is an analgesic, anti-inflammatory, and antipyretic drug with a long duration of action, included in the oxicam subgroup of NSAIDs. Tenoxicam has been studied and found effective for many rheumatic diseases such as rheumatoid arthritis, ankylosing spondylitis, gout, extra-articular disorders, bursitis, tendonitis, and osteoarthritis. The primary aim of this study was to compare the effects of tenoxicam, paracetamol, and tenoxicam-paracetamol combination analgesic applications on the postoperative VAS score of double-jaw surgery patients. The secondary aim was to investigate the effects of these interventions on the number of both opioid and rescue analgesic drug consumption postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-50 aged of both genders who were scheduled for elective bimaxillary surgery
* Classified as American Society of Anesthesiologists (ASA) risk class I or II

Exclusion Criteria:

* having liver or renal dysfunction
* coagulopathy disorder,
* having psychiatric or medical conditions that might impair communication or compliance with the study procedures
* having allergy or contra-indications to the study drugs .pregnancy.
* patients who were planned to undergo additional simultaneous surgical procedures such as genioplasty were not included in the study. -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18-50
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The effects of tenoxicam, paracetamol, and tenoxicam-paracetamol combination on the postoperative 30th minute, first hour and 2th hour VAS (Visual Analog Scale) of double-jaw surgery patients. | at the first hour
  VAS ( Pain intensity was assessed on a 100-mm Visual Analog Scale (VAS), where 0 = no pain and 100 = worst possible pain
The effects of tenoxicam, paracetamol, and tenoxicam-paracetamol combination | at the second hour
  VAS ( Pain intensity was assessed on a 100-mm Visual Analog Scale (VAS), where 0 = no pain and 100 = worst possible pain
The effects of tenoxicam, paracetamol, and tenoxicam-paracetamol combination | at the 24th hour
  VAS ( Pain intensity was assessed on a 100-mm Visual Analog Scale (VAS), where 0 = no pain and 100 = worst possible pain

SECONDARY OUTCOMES:
The secondary efficacy variable was the number of opioid and rescue drug consumptions during the postoperative 24 hours. | during the postoperative 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: seher Orbay Yaşlı, Principal Investigator — Erciyes University Faculty of Dentistry
Locations (1):
- Seher Orbay Yaşlı, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No